CLINICAL TRIAL: NCT03007121
Title: Comparison of Intrathecal Morphine, Epidural Bupivacaine With Sufentanil and Systemic Patient Controlled Analgesia With Morphine for Analgesia After Colorectal Surgery: Prospective Randomised Study.
Brief Title: Intrathecal Morphine Analgesia vs. Continuous Epidural Analgesia vs. Systemic Analgesia in Colorectal Surgery.
Acronym: KOLORIT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Jiri Malek, Assoc. Prof. MD, Ph.D., Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KOLORIT1
Record Dates: First submitted 2016-12-28; First posted 2017-01-02 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Analgesia, Patient-Controlled; Epidural Analgesia; Anesthesia; Spinal; Morphine; Surgery, Colorectal; Intravenous Drug Delivery Systems
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine; Analgesia, Epidural; Sufentanil; Morphine; Analgesia, Patient-Controlled

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Morphine intrathecal (Experimental): An intrathecal administration of preservative-free morphine 0.3 mg in 3 ml NS prepared in a sterile ampoules by a hospital pharmacy will be performed before induction of anaesthesia in a sitting position between L2 and L3 - L4/L5 vertebrae. Standard general anaesthesia will be performed. After surgery, the patients will have the possibility to use PCA device with morphine, bolus dose 1 mg, lock-out interval 5 min for 3 days at a surgical ICU.
  Interventions: Drug: Morphine intrathecal; Drug: Morphine intravenous
- Bupivacaine + Sufentanil epidural (Active Comparator): An epidural catheter will be inserted before induction of anaesthesia in a sitting position between T9 and T10 - T12 and L1 vertebrae. A test dose of 4 ml 0.5 bupivacaine will be administered to rule out intravascular injection or subarachnoid or subdural block. Standard general anaesthesia will be performed. Thirty minutes before the end of the surgery, patients will be administered a bolus of a mixture of bupivacaine 0.5% (3 ml) + sufentanil 10 mcg (2 ml) + NS 5 ml followed by a continuous infusion of a mixture containing in 1 ml bupivacaine 0,125% and sufentanil 0,4 mcg at 8 ml/h. At the same time patients will have the possibility to use PCA device with morphine, bolus dose 1 mg, lock-out interval 5 min for 3 days at a surgical ICU.
  Interventions: Drug: Bupivacaine + Sufentanil epidural; Drug: Morphine intravenous
- Morphine intravenous (Active Comparator): Patients will be administered standard general anaesthesia. After surgery, bolus doses of morphine 2 mg will be administered until level of pain will be < 4 (VAS 0 - 10). Analgesia will be continued by PCA device using morphine, bolus dose 1 mg, lock-out interval 5 min. for 3 days at surgical ICU.
  Interventions: Drug: Morphine intravenous

INTERVENTIONS:
Drug: Morphine intrathecal — Administration of intrathecal injection of 0.3 mg preservative-free morphine in 3 ml NS
  Other Names: Morphine spinal
  Arms: Morphine intrathecal
Drug: Bupivacaine + Sufentanil epidural — Continuous epidural infusion of a mixture containing in 1 ml bupivacaine 0,125% and sufentanil 0,4 mcg at 8 ml/h.
  Other Names: Epidural analgesia with bupivacaine and sufentanil
  Arms: Bupivacaine + Sufentanil epidural
Drug: Morphine intravenous — Patiernt-controlled i.v. analgesia with morphine
  Other Names: Morphine and patient controlled analgesia

SUMMARY:
The purpose of this study is to determine which postoperative analgesia is optimal after colorectal surgery. The investigators will compare intrathecal morphine, continuous epidural analgesia and standard systemic analgesia. All patients will have the possibility to administer themselves intravenous morphine as needed.

DETAILED DESCRIPTION:
Introduction

Colorectal surgery is a frequent operation with expected strong post-operative pain. Thoracic epidural analgesia is a preferred method by many authors, but it is not without risks. As patients in our hospital usually stay at a surgical ICU for 24 hours only and epidural infusion of opioids is prohibited at standard wards according to our hospital standards, it seems to be too demanding method. Systemic analgesia with strong opioids is usually an alternative, but high doses of opioids are known to cause side effects. The last possibility is a single-shot intrathecal injection of morphine which demonstrated long-lasting analgesia after various procedures. The main advantage is easy technique, absence of catheters and low cost. There are not enough studies to decide which method is the most convenient. The purpose of this prospective randomized open clinical study is to determine which postoperative analgesia is optimal after colorectal surgery. The investigators will compare intrathecal morphine, continuous epidural analgesia and compare both methods to standard systemic analgesia. All patients will have the possibility to administer themselves intravenous morphine as needed.

Hypotheses

1. Intrathecal morphine is non-inferior to continuous epidural analgesia
2. ] Intrathecal morphine will decrease the need for i.v. systemic patient controlled analgesia (PCA) with morphine

Aims of the study

Primary aims

1. To demonstrate non-inferiority of analgesia with intrathecal morphine 0.3mg compared to continuous epidural analgesia with 8 ml/hour of mixture of bupivacaine 0.125% and sufentanil 0,4ug/ml. Non-inferiority is defined as consumption of PCA morphine during 24 and 72 hours not higher than 10% compared to control group.
2. To demonstrate significantly lower consumption (at least 10%) of PCA morphine in patients with intrathecal morphine 0.3 mg compared to systemic analgesia with PCA morphine only.

Secondary aims

1. To demonstrate similar or lower side effects of intrathecal morphine compared to epidural or systemic analgesia. The investigators will record number of patients with respiratory rate <8/min, SpO2<90%, changes of blood pressure and pulse rate > 30% above base level before surgery, episodes of postoperative nausea and vomiting
2. To demonstrate the same or shorter interval since surgery to the first bowel movement confirmed by auscultation and interval to the first flatus.
3. To demonstrate the same or lower pain intensity in patients with intrathecal morphine compared to other two groups. The effect will be measured by area below visual analogue scale (0 - 10) pain intensity after 24 and 72 hours

Duration of the study: Three days

Method

Design: Study will be performed as prospective randomized open clinical study

Setting: Surgical ICU

Inclusion criteria: Patients with elective colorectal surgery (left or right hemicolectomy, subtotal colectomy, resection of sigmoid, rectal or cecum)

Exclusion criteria: Known allergy to any of drugs used, coagulopathy, sepsis, cognitive dysfunction and/or inability to understand instruction. Pregnancy (is assessed as a part of pre-operative examination). Abuse of drugs or administration of morphine therapy 5 or less days before surgery. Idiopathic bowel disease.

Anesthesia: General anesthesia will be performed in all groups using propofol for induction and rocuronium for intubation and muscle relaxation. Patients will be ventilated to normocapnia by oxygen + air + desflurane mixture. Sufentanil 5 - 10 mcg will be administered if needed. Paracetamol 1 g i.v. will be administered approximately 30 min before the end of anesthesia and ondansetron 4 mg i.v. will be administered 10 min. before the end of anesthesia. At the end of anesthesia patients will be administered atropine and neostigmine to obtain TOF ration >90%.

Standard postoperative analgesia: All patients will be administered paracetamol 1g i.v. every 6 h for next 72 hours and can use PCA morphine, bolus dose 1 mg, lock-out interval 5 min. for 3 days at surgical ICU.

Monitoring: Except of standard anesthesia and ICU monitoring (ECG, pulse oximetry and non-invasive blood pressure) pain intensity (VAS 0 - 10) and side effects (see above) will be recorded.

Power analysis: Total number of patients to demonstrate primary aims is 75 divided in ratio 1:2:2; n=15 in systemic analgesia group (PCA) and n=30 in each group with epidural and intrathecal analgesia. Standard tests will be used to analyse results. P value < 0.05 will be considered significant.

Interventions:

1. Systemic analgesia: Patients will be administered standard general anesthesia. After surgery, bolus doses of morphine 2 mg will be administered until level of pain will be < 4 (VAS 0 - 10). Analgesia will be continued by PCA device using morphine, bolus dose 1 mg, lock-out interval 5 min. for 3 days at surgical ICU.
2. Epidural analgesia: An epidural catheter will be inserted before induction of anesthesia in a sitting position between T9 and T10 - T12 and L1 vertebrae. A test dose of 4 ml 0.5 bupivacaine will be administered to rule out intravascular injection or subarachnoid or subdural block. Standard general anesthesia will be performed. Thirty minutes before the end of the surgery, patients will be administered a bolus of a mixture of bupivacaine 0.5% (3 ml) + sufentanil 10 mcg (2 ml) + NS 5 ml followed by a continuous infusion of a mixture containing in 1 ml bupivacaine 0.125% and sufentanil 0.4 mcg at 8 ml/h. At the same time patients will have the possibility to use PCA device with morphine, bolus dose 1 mg, lock-out interval 5 min for 3 days at a surgical ICU. Epidural infusion will be stopped 24 hours after surgery.
3. Intrathecal analgesia: An intrathecal administration of preservative-free morphine 0.3 mg in 3 ml NS prepared in sterile ampoules by a hospital pharmacy will be performed before induction of anesthesia in a sitting position between L2 and L3 - L4/L5 vertebrae. Standard general anesthesia will be performed. After surgery, the patients will have the possibility to use PCA device with morphine, bolus dose 1 mg, lock-out interval 5 min for 3 days at a surgical ICU.

ELIGIBILITY:
Inclusion Criteria:

* Patients with elective colorectal surgery (left or right hemicolectomy, subtotal colectomy, resection of sigmoid, rectal or cecum)

Exclusion Criteria:

* Known allergy to any of drugs used, coagulopathy, sepsis, cognitive dysfunction and/or inability to understand instruction.
* Pregnancy (is assessed as a part of pre-operative examination).
* Abuse of drugs or morphine therapy before surgery.
* Idiopathic bowel disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
Non-inferiority of analgesia with intrathecal morphine 0.3mg compared with epidural mixture bupivacaine 0.125% and sufentanil 0,4ug/ml. | Within the first 3 days after surgery
  Non-interiority is defined as difference in morphine consumption during patient-controlled analgesia no more than 10%
Better analgesia after intrathecal morphine compared to systemic analgesia with morphine | Within the first 3 days after surgery
  Lower consumption of PCA morphine in patients with intrathecal morphine compared to systemic analgesia with PCA morphine only.

SECONDARY OUTCOMES:
Side effects of intrathecal morphine compared to epidural or systemic analgesia | Within the first 3 days after surgery
  Number of patients with respiratory rate <8/min, SpO2<90%, changes of blood pressure and pulse rate > 30% above base level before surgery, episodes of postoperative nausea and vomiting, interval since surgery to the first bowel movement confirmed by auscultation and interval to the first flatus.
Pain intensity | Within the first 3 days after surgery
  Area below visual analogue scale (0 - 10) pain intensity after 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jiri Malek, M.D., Principal Investigator — 3rd Medical Faculty, Charles University and University Hiospital Kralovske Vinohrady
Locations (1):
- University Hospital Kralovske Vinohrady, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Devys JM, Mora A, Plaud B, Jayr C, Laplanche A, Raynard B, Lasser P, Debaene B. Intrathecal + PCA morphine improves analgesia during the first 24 hr after major abdominal surgery compared to PCA alone. Can J Anaesth. 2003 Apr;50(4):355-61. doi: 10.1007/BF03021032. English, French. PMID 12670812
- [Background] Beaussier M, Weickmans H, Parc Y, Delpierre E, Camus Y, Funck-Brentano C, Schiffer E, Delva E, Lienhart A. Postoperative analgesia and recovery course after major colorectal surgery in elderly patients: a randomized comparison between intrathecal morphine and intravenous PCA morphine. Reg Anesth Pain Med. 2006 Nov-Dec;31(6):531-8. doi: 10.1016/j.rapm.2006.06.250. PMID 17138196
- [Background] Sakowska M, Docherty E, Linscott D, Connor S. A change in practice from epidural to intrathecal morphine analgesia for hepato-pancreato-biliary surgery. World J Surg. 2009 Sep;33(9):1802-8. doi: 10.1007/s00268-009-0131-2. PMID 19548026
- [Background] Virlos I, Clements D, Beynon J, Ratnalikar V, Khot U. Short-term outcomes with intrathecal versus epidural analgesia in laparoscopic colorectal surgery. Br J Surg. 2010 Sep;97(9):1401-6. doi: 10.1002/bjs.7127. PMID 20603849
- [Background] Levy BF, Scott MJ, Fawcett W, Fry C, Rockall TA. Randomized clinical trial of epidural, spinal or patient-controlled analgesia for patients undergoing laparoscopic colorectal surgery. Br J Surg. 2011 Aug;98(8):1068-78. doi: 10.1002/bjs.7545. Epub 2011 May 17. PMID 21590762
- [Background] Werawatganon T, Charuluxananan S. WITHDRAWN: Patient controlled intravenous opioid analgesia versus continuous epidural analgesia for pain after intra-abdominal surgery. Cochrane Database Syst Rev. 2013 Mar 28;2013(3):CD004088. doi: 10.1002/14651858.CD004088.pub3. PMID 23543529
- [Background] Rodgers A, Walker N, Schug S, McKee A, Kehlet H, van Zundert A, Sage D, Futter M, Saville G, Clark T, MacMahon S. Reduction of postoperative mortality and morbidity with epidural or spinal anaesthesia: results from overview of randomised trials. BMJ. 2000 Dec 16;321(7275):1493. doi: 10.1136/bmj.321.7275.1493. PMID 11118174
- [Background] Rigg JR, Jamrozik K, Myles PS, Silbert BS, Peyton PJ, Parsons RW, Collins KS; MASTER Anaethesia Trial Study Group. Epidural anaesthesia and analgesia and outcome of major surgery: a randomised trial. Lancet. 2002 Apr 13;359(9314):1276-82. doi: 10.1016/S0140-6736(02)08266-1. PMID 11965272
- [Background] Manion SC, Brennan TJ. Thoracic epidural analgesia and acute pain management. Anesthesiology. 2011 Jul;115(1):181-8. doi: 10.1097/ALN.0b013e318220847c. No abstract available. PMID 21606825
- [Background] Moen V, Dahlgren N, Irestedt L. Severe neurological complications after central neuraxial blockades in Sweden 1990-1999. Anesthesiology. 2004 Oct;101(4):950-9. doi: 10.1097/00000542-200410000-00021. PMID 15448529
- [Background] Meylan N, Elia N, Lysakowski C, Tramer MR. Benefit and risk of intrathecal morphine without local anaesthetic in patients undergoing major surgery: meta-analysis of randomized trials. Br J Anaesth. 2009 Feb;102(2):156-67. doi: 10.1093/bja/aen368. PMID 19151046
- [Background] De Pietri L, Siniscalchi A, Reggiani A, Masetti M, Begliomini B, Gazzi M, Gerunda GE, Pasetto A. The use of intrathecal morphine for postoperative pain relief after liver resection: a comparison with epidural analgesia. Anesth Analg. 2006 Apr;102(4):1157-63. doi: 10.1213/01.ane.0000198567.85040.ce. PMID 16551916
- [Background] Holte K, Kehlet H. Epidural analgesia and risk of anastomotic leakage. Reg Anesth Pain Med. 2001 Mar-Apr;26(2):111-7. doi: 10.1053/rapm.2001.21241. PMID 11251133